CLINICAL TRIAL: NCT00002687
Title: Phase 1 Trial of Subcutaneous [SC]; Outpatient Interleukin-2 for Patients With Advanced Mycosis Fungoides [Stage IIb, III, IV]
Brief Title: Interleukin-2 in Treating Patients With Mycosis Fungoides
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000064412; UW-24218-A/E; NCI-V95-0758
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-11

CONDITIONS: Lymphoma
Keywords: stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome
MeSH Terms: conditions — Lymphoma; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — aldesleukin

INTERVENTIONS:
Biological: aldesleukin

SUMMARY:
RATIONALE: Interleukin-2 may stimulate a person's white blood cells to kill cancer cells.

PURPOSE: Phase I trial to study the effectiveness of interleukin-2 in treating patients who have mycosis fungoides.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and toxicity of interleukin-2 in patients with stage IIB-IV mycosis fungoides.
* Determine the response rate of patients treated with this regimen.
* Determine the immunologic response to this regimen in peripheral blood leukocytes and serum of these patients.

OUTLINE: This is a dose escalation study.

Patients receive interleukin-2 (IL-2) subcutaneously on days 1-5 during weeks 1-3 and on days 1-3 and 5 during week 4. Treatment repeats every 4 weeks for 4 courses.

Cohorts of 3-6 patients receive escalating doses of IL-2 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 3 of 6 patients experience dose-limiting toxicity. Six additional patients receive IL-2 at 1 dose level preceding the MTD.

Patients are followed at least 3 times during year 1 and then annually thereafter.

PROJECTED ACCRUAL: A total of 16-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Clinically and histologically proven diagnosis of 1 of the following:

  * Mycosis fungoides (MF) meeting 1 of the following conditions:

    * Stage IIB disease that has failed psoralen ultraviolet A (PUVA) light therapy and topical chemotherapy (mechlorethamine and/or carmustine)
    * Stage III disease with generalized erythroderma
    * Stage IV disease with biopsy proven nodal or visceral involvement
  * Sezary syndrome

    * Stage III MF with a minimum of 20% Sezary cells (based on total WBC)
* No clinically significant ascites or pleural effusion

  * Clinically significant pleural effusion defined as shortness of breath with oxygen saturation less than 90%

PATIENT CHARACTERISTICS:

Age:

* 18 to 80

Performance status:

* Karnofsky 70-100%

Life expectancy:

* At least 16 weeks

Hematopoietic:

* See Disease Characteristics
* WBC at least 3,500/mm^3
* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 11.5 g/dL

Hepatic:

* Bilirubin less than 2.5 times normal
* SGOT less than 2.5 times normal

Renal:

* Creatinine no greater than 2.0 mg/dL
* No nephrotic syndrome

Cardiovascular:

* No history of myocardial infarction or congestive heart failure
* No symptomatic coronary artery disease
* No clinically manifest hypotension
* No severe hypertension
* No arrhythmia on electrocardiogram
* No edema
* No contraindication to pressor agents

Pulmonary:

* See Disease Characteristics
* No dyspnea at rest or severe exertional dyspnea

Neurologic:

* No significant CNS dysfunction, including any of the following:

  * Seizure disorder
  * Active cerebrovascular disease
  * Dementia or delirium

Other:

* No autoimmune disease, including psoriasis
* No uncontrolled peptic ulcer disease
* No uncontrolled infection
* No history of adverse reaction to interleukin-2
* HIV and HTLV-I negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior systemic or topical chemotherapy (6 weeks since prior mitomycin or nitrosoureas)

Endocrine therapy:

* At least 1 week since prior corticosteroids
* No concurrent corticosteroids

Radiotherapy:

* At least 4 weeks since prior radiotherapy

Surgery:

* No prior organ allograft
* At least 3 weeks since other prior major surgery

Other:

* At least 4 weeks since prior immunosuppressive therapy
* At least 2 weeks since prior phototherapy (ultraviolet B [UVB] or PUVA light therapy)
* No concurrent phototherapy (UVB or PUVA light therapy)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1995-02; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A. Thompson, MD, Study Chair — Seattle Cancer Care Alliance
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States